CLINICAL TRIAL: NCT04995094
Title: A Phase II, Neoadjuvant, Randomized, Multicenter Study of Imprime PGG Plus Pembrolizumab in Subjects With Stage III, Resectable Melanoma
Brief Title: Study of Neoadjuvant Imprime PGG and Pembrolizumab for Stage III, Resectable Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges, study not feasible
Sponsor: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGG-MEL2021
Record Dates: First submitted 2021-07-19; First posted 2021-08-06 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Pathologic Stage III Cutaneous Melanoma AJCC v8
Keywords: Stage III; resectable; melanoma; Imprime; Imprime PGG; pembrolizumab; neoadjuvant
MeSH Terms: conditions — Melanoma | interventions — BTH1677; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Randomized
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imprime PGG + Pembrolizumab (Investigational ARM) (Experimental): Imprime PGG + Pembrolizumab (Investigational ARM)
  Interventions: Biological: Imprime PGG; Biological: Pembrolizumab
- Pembrolizumab (Control ARM) (Active Comparator): Pembrolizumab (Control ARM)
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Imprime PGG — Imprime PGG is a soluble, β-1,3/1,6 glucan isolated from the cell wall of a proprietary Saccharomyces cerevisiae yeast strain. Imprime PGG acts as a Pathogen-Associated Molecular Pattern (PAMP). Imprime will be administered at a dose of 4 mg/kg IV over a 2-hour infusion time on Days 1, 8 and 15 of each 3-week treatment cycle.
  Other Names: BTH1677
  Arms: Imprime PGG + Pembrolizumab (Investigational ARM)
Biological: Pembrolizumab — Pembrolizumab is a humanized monoclonal antibody against the programmed death receptor-1 (PD-1) protein. Pembrolizumab will be administered at 200 mg IV Q3W for 9 weeks.
  Other Names: KEYTRUDA®

SUMMARY:
Approximately 50 ABA+ subjects with resectable, Stage III (IIIB, IIIC, or IIID) melanoma will be included in the study and randomized in a 3:2 ratio to neoadjuvant treatment with Imprime PGG plus pembrolizumab vs. pembrolizumab monotherapy. A baseline, reference biopsy and a PET/CT scan will be obtained prior to commencing 3 cycles (9 weeks) of neoadjuvant treatment with either regimen. During Week 5, subjects will provide another biopsy to assess treatment effects on the tumor and its microenvironment. At the completion of neoadjuvant treatment and before surgery, subjects will undergo another PET/CT scan to assess radiological and metabolic response compared to baseline.

DETAILED DESCRIPTION:
Approximately 50 ABA+ subjects with resectable, Stage III (IIIB, IIIC, or IIID) melanoma will be included in the study and randomized in a 3:2 ratio to neoadjuvant treatment with Imprime PGG plus pembrolizumab vs. pembrolizumab monotherapy. A baseline, reference biopsy and a PET/CT scan will be obtained prior to commencing 3 cycles (9 weeks) of neoadjuvant treatment with either regimen. During Week 5, subjects will provide another biopsy to assess treatment effects on the tumor and its microenvironment. At the completion of neoadjuvant treatment and before surgery, subjects will undergo another PET/CT scan to assess radiological and metabolic response compared to baseline.

Subjects will then undergo surgical resection. A pre-surgical assessment of operability will be done by the responsible surgeon, and the investigator will ensure that adverse events occurring during the treatment period have resolved to the minimal acceptable level that would not place the subject at undue risk or delay surgery for more than 1 week after the last dose of Imprime or 3 weeks after last dose of pembrolizumab, when subjects will undergo surgical resection.

The surgical specimen will be locally and centrally assessed by a pathologist to determine the pathological response (pCR, pMR, pPR) induced by the neoadjuvant treatment (central read will be blinded). Following surgery, subjects will be followed for safety for 90 days. The total duration of systemic treatment will be 3 cycles (9 weeks). In the Investigational arm, surgery should be performed no more than a week after the subject's last dose of Imprime PGG and in the Control arm, surgery should be performed within 3 weeks of the subject's last dose of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. ≥18 years of age
3. Histologically confirmed diagnosis of resectable* AJCC (8th edition) Stage IIIB, IIIC or IIID cutaneous or unknown primary melanoma (except for any in-transit or satellite metastases) (*Resectable Stage III disease is defined as disease that is amenable to complete tumor resection (anticipated to be an R0 resection) as judged as judged by the responsible surgeon. Criteria to judge resectability include, but are not limited to, lesions located in anatomically inaccessible areas, or invading vascular or neural structures, or technical or other reasons preventing their complete removal)
4. No prior systemic treatment for melanoma (subjects who were previously resected, relapsed and are once again resectable are eligible)
5. RECIST 1.1 measurable disease:

   a.) ≥ 10mm in the longest diameter for primary (if applicable) lesions or lymph node and/or ≥ 15mm in the shortest diameter for lymph nodes b) Sufficient nodal +/1 primary lesions amenable to ≥ 2 excisional/ core biopsies
6. No prior radiotherapy to nodal basin
7. Subject consents to provide 2 newly obtained core or excisional biopsies from non-nodal, non-bone lesions (within 28 days prior to C1D1 and during Wk 5 of treatment), the use of the resected surgical specimen and additional blood samples for translational research correlative studies
8. Have peripheral blood levels of IgG anti-β-glucan antibody (ABA) of ≥ 20 mcg/mL as determined by an ELISA test prior to (within 90 days) start of study treatment
9. ECOG PS 0-1 (within 7 days of starting treatment)
10. Estimated life expectancy of ≥12 weeks, in the opinion of the Investigator
11. Adequate organ function, including all of the following within 15 days before Day 1:

    a.) Hematological: i.) Absolute neutrophil count (ANC) ≥ 1.5×109/L (> 1,500/mm3) (subject may not use G-CSF or GM-CSF to achieve this level) ii.) Platelets ≥ 100×109/L (>100,000 per mm3) iii.) Hemoglobin level >9 gm/dL. Packed red blood cell transfusion is acceptable, as long as the subject has a stable result of >9 gm/dL for at least 1week post-transfusion. Erythropoietin should not be used to achieve this level iv.) Adequate coagulation function at screening as determined by prothrombin time (PT) International Normalized Ratio (INR) < 1.5 times the upper limit of normal (ULN) and partial thromboplastin time (PTT) < 1.5 times the ULN v.) Lymphocyte count >1500 cells/mL b.) Intact immune system as demonstrated by CD4 count >500 cells/mm3 and CD8 count >150 cells/mm3 c.) Renal: i.) Serum creatine or measured and calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN and creatinine clearance ≥30 mL/min, per Cockcroft Gault formula d.) Hepatic: i.) Serum total bilirubin ≤1.5× ULN or direct bilirubin ≤ ULN for a subject with total bilirubin levels >1.5× ULN ii.) AST/ALT < 2.5 x ULN iii.) Albumin >3 g/dL
12. Have a negative PCR test at screening for SARS-COV-2 RNA
13. Women of childbearing potential (WOCBP) must have 2 negative serum or urine pregnancy tests during Screening, the second within 24 hours prior to the first administration of study drug, and must agree to use highly effective physician-approved contraception from Screening to a minimum of 90 days following the last study drug administration
14. Willing and able to comply with all protocol-specified assessments and the study visit schedule.

Exclusion Criteria:

1. Prior therapy for melanoma (resection of a previous melanoma lesion is acceptable)
2. Subjects with uveal or mucosal melanoma
3. Pregnant, lactating or not practicing adequate contraception (premenopausal women), or expecting to conceive or father children within the duration of the trial, starting from Screening to 90 days following the last dose of drug administration
4. Prior radiotherapy in the previous 2 weeks. Radiotherapy to presenting tumor is prohibited
5. Administration of a live, attenuated vaccine within 28 days prior to Day 1 or anticipation that such a live attenuated vaccine will be required during the study
6. History of autoimmune disease, including but not limited to inflammatory bowel disease, systemic lupus erythematosus, and autoimmune hepatitis, requiring systemic treatment in previous 12 months
7. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone [>10mg], dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 15 days prior to Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial
8. Immunodeficiency, natural or iatrogenic (steroids, immunosuppressants)
9. History of malignancy within the last 3 years. Subjects with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Subjects with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years
10. Known CNS metastasis of leptomeningeal disease
11. Known history of HIV, Hepatitis B, active Hepatitis C or tuberculosis
12. History of pneumonitis including interstitial lung disease
13. Has a known hypersensitivity to any component of protocol therapy, or their vehicle(s)
14. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (NYHA Grade 2), unstable angina pectoris, cardiac arrhythmia, any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification or psychiatric illness
15. Has a fever >38oC within 3 days before the first dose of study treatment
16. Had previous exposure to Imprime PGG
17. Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF, or recombinant erythropoietin) within 4 weeks prior to Study Day 1
18. Any condition which could interfere with, or the treatment for which might interfere with the conduct of the study or which would, in the opinion of the Investigator, unacceptably increase the subject's risk by participating in the study
19. Subject is under legal custodianship
20. First-degree relatives of the investigator, study staff or the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-02-18 (Estimated); Study Completion 2023-05-18 (Estimated)

PRIMARY OUTCOMES:
Pathological Response Rate (pRR) | Within 18 months of last patient enrolled
  To determine the pathological response rate (pRR) in the surgically resected specimen post completion of neoadjuvant therapy with Imprime PGG plus pembrolizumab vs pembrolizumab monotherapy

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Within 24 months of last patient enrolled
  Radiological overall response rate (ORR) (by RECIST 1.1)
Incidence of Treatment-Emergent Adverse Events | Within 24 months of last patient enrolled
  Safety of neoadjuvant treatment (incidence of treatment-emergent adverse events, change from baseline in physical findings, ECGs, and laboratory results)
Metabolic Response Rate | Within 24 months of last patient enrolled
  Metabolic Response Rate (assessed by PET per EORTC recommendations)
Correlation of Metabolic Response Rate (pathological response) | Within 24 months of last patient enrolled
  Correlation of metabolic response rate with pathological response
Correlation of metabolic Response Rate (RECIST response) | Within 24 months of last patient enrolled
  Correlation of metabolic response rate with RECIST response.
Correlation of Pathological Response Rate (RECIST) | Within 24 months of last patient enrolled
  Correlation of pathological response rate with RECIST response
Incidence of Surgical Delays or Complications | Within 24 months of last patient enrolled
  Incidence of surgical delays or complications, including post-operative infections
Opinion of Operability | Within 24 months of last patient enrolled
  Comparison pre and post treatment portion of participants with disease amendable to complete tumor resection as judged by the responsible surgeon to compare surgeon's opinion of operability
Severity of treatment-emergent adverse events | Within 24 months of last patient enrolled
  Safety of neoadjuvant treatment (treatment-emergent adverse events, change from baseline in physical findings, ECGs, and laboratory results)

OTHER OUTCOMES:
Circulating Tumor DNA (ctDNA) | Within 24 months of last patient enrolled
  Measurement of circulating tumor DNA (ctDNA)
Degree of Necrosis and Genetic Markers in Tumor Tissue | Within 24 months of last patient enrolled
  Measurement of degree of necrosis and genetic markers in tumor tissue
Tumor Microenvironment (TME) | Within 24 months of last patient enrolled
  Assessment of tumor microenvironment (TME) composition in biopsies at baseline and mid-treatment (during Wk 5), and a surgical resection specimen
Measurement of Immune Cell Populations (peripheral blood) | Within 24 months of last patient enrolled
  Measurement of pre and post treatment of immune cell populations in peripheral blood
Cytokine Profiles (peripheral blood) | Within 24 months of last patient enrolled
  Assessment of cytokine profiles in peripheral blood before and during treatment
Correlation of Anti-beta Glucan Antibody (ABA) | Within 24 months of last patient enrolled
  Correlation of anti-beta glucan antibody (ABA) expression levels with pathological, clinical & translational outcomes

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Innovative Clinical Research Institute, Whittier, California
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Allegheny Health Network, Pittsburgh, Pennsylvania